CLINICAL TRIAL: NCT03834844
Title: Mindfulness Meditation and Patient Education for Symptom Management in Individuals With Atrial Fibrillation(AF): Do They Need to Be Offered Together?
Brief Title: Meditation and Education That is Nurse Delivered for Symptom Management in Paroxysmal Atrial Fibrillation (PAF)
Acronym: MEND-AF2
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Paul Wang, Professor of Medicine, Stanford University
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: IRB-44919
Record Dates: First submitted 2019-02-06; First posted 2019-02-08 (Actual); Last update posted 2024-12-02 (Actual); Status verified 2024-11

CONDITIONS: Paroxysmal Atrial Fibrillation
Keywords: Symptom Management; Quality of Life; Anxiety
MeSH Terms: conditions — Atrial Fibrillation; Anxiety Disorders | interventions — Meditation

STUDY DESIGN:
Intervention Model Description: 2 x 2 factorial design
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (8):
- Usual Care (No Intervention): patient receives same care as patients not enrolled in study intervention
- AF education (Experimental): Participant receives 6 modules of AF education topics that are intended to be completed consecutively, one each week.
  Interventions: Other: AF Education
- Mindfulness Meditation Practice (Experimental): Each participant watches an mindfulness meditation introductory video in the initial session and then is asked to practice for 10 minutes each day using a guided audio, which includes a different topic each week. The time duration of the guided meditations increases to 15 minutes each day during Weeks 3-6.
  Interventions: Behavioral: Meditation
- Weekly Phone Calls (Experimental): Each week for the six-week intervention, the researcher will contact the participant by phone at an agreed upon time and will discuss any questions, issues or concerns that are voiced by the participant within 5-15 minutes.
  Interventions: Other: Phone Calls
- AF Education and Mindfulness Meditation (Experimental): Participant receives 6 modules of AF education topics that are intended to be completed consecutively, one each week. Each participant watches an mindfulness meditation introductory video in the initial session and then is asked to practice for 10 minutes each day using a guided audio, which includes a different topic each week. The time duration of the guided meditations increases to 15 minutes each day during Weeks 3-6.
  Interventions: Behavioral: Meditation; Other: AF Education
- AF Education and Weekly Phone Calls (Experimental): Participant receives 6 modules of AF education topics that are intended to be completed consecutively, one each week. Each week for the six-week intervention, the researcher will contact the participant by phone at an agreed upon time and will discuss any questions, issues or concerns that are voiced by the participant within 5-15 minutes.
  Interventions: Other: AF Education; Other: Phone Calls
- Mindfulness Meditation and Phone Calls (Experimental): Each participant watches an mindfulness meditation introductory video in the initial session and then is asked to practice for 10 minutes each day using a guided audio, which includes a different topic each week. The time duration of the guided meditations increases to 15 minutes each day during Weeks 3-6. Each week for the six-week intervention, the researcher will contact the participant by phone at an agreed upon time and will discuss any questions, issues or concerns that are voiced by the participant within 5-15 minutes.
  Interventions: Behavioral: Meditation; Other: Phone Calls
- Meditation and Education and Phone Calls (Experimental): Each participant watches an mindfulness meditation introductory video in the initial session and then is asked to practice for 10 minutes each day using a guided audio, which includes a different topic each week. Participant receives 6 modules of AF education topics that are intended to be completed consecutively, one each week. The time duration of the guided meditations increases to 15 minutes each day during Weeks 3-6. Each week for the six-week intervention, the researcher will contact the participant by phone at an agreed upon time and will discuss any questions, issues or concerns that are voiced by the participant within 5-15 minutes.
  Interventions: Behavioral: Meditation; Other: AF Education; Other: Phone Calls

INTERVENTIONS:
Behavioral: Meditation — Guided Meditation for 10-15 minutes daily for 6 days/week for 6 weeks
  Arms: AF Education and Mindfulness Meditation; Meditation and Education and Phone Calls; Mindfulness Meditation Practice; Mindfulness Meditation and Phone Calls
Other: AF Education — 6 weekly education modules on topics related to AF
  Arms: AF Education and Mindfulness Meditation; AF Education and Weekly Phone Calls; AF education; Meditation and Education and Phone Calls
Other: Phone Calls — Weekly phone call to discuss patient concerns or questions
  Arms: AF Education and Weekly Phone Calls; Meditation and Education and Phone Calls; Mindfulness Meditation and Phone Calls; Weekly Phone Calls

SUMMARY:
The aim of this project is to determine whether the entire intervention (Mindfulness meditation, AF education, and weekly phone visits) that is nurse delivered to individuals with paroxysmal atrial fibrillation is more effective than a combination, single or no intervention in the reduction of overall AF symptoms, anxiety, and negative illness perception; or the improvement of quality of life (QOL) and functional status.

ELIGIBILITY:
Inclusion Criteria:

1. Individuals with Symptomatic Paroxysmal Atrial Fibrillation
2. A symptomatic episode of PAF within last 6 months
3. 18 years old or greater
4. Able to read and understand English
5. Able to participate in weekly phone calls
6. Able to attend two video visit/phone sessions that are 6 weeks apart

Exclusion Criteria:

1. Diagnosed with low cardiac function (NYHA Class IV)
2. Life expectancy of less than 6 months
3. Hospitalized in prior 3 months for illness other than PAF
4. Previously practiced mindfulness
5. Cognitive impairment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — All
Enrollment: 50 (Actual)
Dates: Start 2018-05-01 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline Atrial Fibrillation Symptom Burden and Symptom Severity Scores | Baseline (Initial), Post-Intervention (6 weeks)
  Atrial Fibrillation Burden and Symptom Severity will be calculated from the patient-completed responses on the Atrial Fibrillation Symptom Severity Scale-Symptom Burden can range from 3.25 (minimally bothersome) to 30 (continuous symptomatic episodes) and is based on event frequency (1-10), duration (1.25-10), and global episode (1-10). Symptom severity is based on symptom specific subscale with range from 0(no symptoms) to 35 (severe symptoms).
Change from Baseline Atrial Fibrillation Symptom Burden and Symptom Severity Scores | Baseline (Initial), 6 month
  Atrial Fibrillation Burden and Symptom Severity will be calculated from the patient-completed responses on the Atrial Fibrillation Symptom Severity Scale-Symptom Burden can range from 3.25 (minimally bothersome) to 30 (continuous symptomatic episodes) and is based on event frequency (1-10), duration (1.25-10), and global episode (1-10). Symptom severity is based on symptom specific subscale with range from 0(no symptoms) to 35 (severe symptoms).
Change from Baseline Atrial Fibrillation Symptom Burden and Symptom Severity Scores | Baseline (Initial), 12 month
  Atrial Fibrillation Burden and Symptom Severity will be calculated from the patient-completed responses on the Atrial Fibrillation Symptom Severity Scale-Symptom Burden can range from 3.25 (minimally bothersome) to 30 (continuous symptomatic episodes) and is based on event frequency (1-10), duration (1.25-10), and global episode (1-10). Symptom severity is based on symptom specific subscale with range from 0(no symptoms) to 35 (severe symptoms).
Change from Baseline in AF Quality of Life Score | Baseline (Initial), Post-Intervention (6 weeks)
  Quality of Life will be assessed using a patient completed questionnaire, Atrial Fibrillation Effect on Quality of Life Questionnaire. The AFEQT score is a combined score of 21 items (21-100) with a higher score representing greater QOL.
Change from Baseline in AF Quality of Life Score | Baseline (Initial), 6 month
  Quality of Life will be assessed using a patient completed questionnaire, Atrial Fibrillation Effect on Quality of Life Questionnaire. The AFEQT score is a combined score of 21 items (21-100) with a higher score representing greater QOL.
Change from Baseline in AF Quality of Life Score | Baseline (Initial), 12 month
  Quality of Life will be assessed using a patient completed questionnaire, Atrial Fibrillation Effect on Quality of Life Questionnaire. The AFEQT score is a combined score of 21 items (21-100) with a higher score representing greater QOL.

SECONDARY OUTCOMES:
Change from Baseline in Anxiety | Baseline (Initial), Post-Intervention (6 weeks)
  Anxiety will be measured using the Cardiac Anxiety Questionnaire with a calculated score (0-72) and higher scores indicate greater heart focused anxiety.
Change from Baseline in Anxiety | Baseline (Initial), 6 months
  Anxiety will be measured using the Cardiac Anxiety Questionnaire with a calculated score (0-72) and higher scores indicate greater heart focused anxiety.
Change from Baseline in Anxiety | Baseline (Initial), 12 months
  Anxiety will be measured using the Cardiac Anxiety Questionnaire with a calculated score (0-72) and higher scores indicate greater heart focused anxiety.

CONTACTS AND LOCATIONS:
Overall Officials: Linda Ottoboni, PhD, Principal Investigator — Clinician and research scientist
Locations (1):
- Stanford Health Care, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: No